CLINICAL TRIAL: NCT01869036
Title: Use of Caudal Anesthesia Supplemented With Morphine in Children Undergoing Renal Surgery - Prospective Study
Brief Title: Use of Caudal Anesthesia Supplemented With Morphine in Children Undergoing Renal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 82/12
Record Dates: First submitted 2012-08-07; First posted 2013-06-05 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Anesthesia, Caudal
Keywords: Caudal; anesthesia; morphine; children
MeSH Terms: interventions — Anesthesia, Caudal; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- caudal anesthesia (Active Comparator)
  Interventions: Drug: caudal anesthesia
- caudal anesthesia supplemented with morphine (Active Comparator)
  Interventions: Drug: caudal anesthesia supplemented with morphine

INTERVENTIONS:
Drug: caudal anesthesia — Standard caudal anesthesia (Marcaine 2mg/kg)
  Other Names: sacral epidural anesthesia
  Arms: caudal anesthesia
Drug: caudal anesthesia supplemented with morphine — Caudal anesthesia supplemented with Morphine (10 µg/kg in children less than 10 kg and 20 µg/kg in children more than 10 kg)
  Arms: caudal anesthesia supplemented with morphine

SUMMARY:
The aim of this study is to test an efficacy and safety of supplemented by Morphine caudal anesthesia in children who undergo renal surgery in our department.

DETAILED DESCRIPTION:
The kidney surgery is a significant part of surgical armamentarium in pediatric urology. The common operations are open and laparoscopic pyeloplasty, partial nephrectomy open and laparoscopic and laparoscopic nephrectomy.

One of the main goals in the postoperative period is to provide a painless recovery following by early mobilization of the child and early discharge home. Caudal anesthesia has become a gold standard in the renal surgery providing painless postoperative period, allowing earlier child feeding and speedy recovery. However some researchers have pointed out that caudal anesthesia with supplemented with Marcaine may provide painless postoperative period only for a very limited period of time and required additional painkiller therapy during postoperative period. Caudal anesthesia supplemented with Morphine has demonstrated their benefits in children who undergo infraumbilical surgery.

ELIGIBILITY:
Inclusion Criteria:

* children who are scheduled for renal surgery from two months age to puberty
* operations are open and laparoscopic pyeloplasty, partial nephrectomy open and laparoscopic and laparoscopic nephrectomy

Exclusion Criteria:

* malignancy

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
statistical diffirence in intraoperative and postoperative narcotic requirements + filling of the pain assessment questionnaire | at the end of operation (anesthesiological report) and at the end of 1 post-op day (nurse report)
  The following parameters will be compared between two groups: the length of surgery, intraoperative and postoperative narcotic requirements. The children parents or children thyself will be asked to fill out the pain assessment questionnaire.

SECONDARY OUTCOMES:
Side-effects measuring | during operation and within 1 post-op day
  Side-effects such as vomiting, itching, respiratory depression, hypotension, and bradycardia will be observed. Oral intake and discharge home will be recorded. Complications rate will be recorded and compared between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Chertin, MD, Principal Investigator — Head, The Department of Pediatric Urology, Shaare Zedek Medical Center, Clinical Professor in Surgery/Urology, Faculty of Medicine, Hebrew University, Jerusalem, Israel
Locations (1):
- The Department of Pediatric Urology, Shaare Zedek Medical Center, Faculty of Medicine, Hebrew University, Jerusalem, Israel

REFERENCES:
- [Background] Mayhew JF, Brodsky RC, Blakey D, Petersen W. Low-dose caudal morphine for postoperative analgesia in infants and children: a report of 500 cases. J Clin Anesth. 1995 Dec;7(8):640-2. doi: 10.1016/0952-8180(95)00089-5. PMID 8747562
- [Background] Fernandes ML, Pires KC, Tiburcio MA, Gomez RS. Caudal bupivacaine supplemented with morphine or clonidine, or supplemented with morphine plus clonidine in children undergoing infra-umbilical urological and genital procedures: a prospective, randomized and double-blind study. J Anesth. 2012 Apr;26(2):213-8. doi: 10.1007/s00540-011-1297-y. Epub 2011 Dec 10. PMID 22159880
- [Background] Singh R, Kumar N, Singh P. Randomized controlled trial comparing morphine or clonidine with bupivacaine for caudal analgesia in children undergoing upper abdominal surgery. Br J Anaesth. 2011 Jan;106(1):96-100. doi: 10.1093/bja/aeq274. Epub 2010 Oct 14. PMID 20952427
- [Background] Cesur M, Alici HA, Erdem AF, Yapanoglu T, Silbir F. Effects of reduction of the caudal morphine dose in paediatric circumcision on quality of postoperative analgesia and morphine-related side-effects. Anaesth Intensive Care. 2007 Oct;35(5):743-7. doi: 10.1177/0310057X0703500514. PMID 17933162